CLINICAL TRIAL: NCT01784692
Title: Pilot Study to Evaluate Immunopotentiating Effects of Immulina in Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Gailen D. Marshall, Professor of Medicine and Pediatrics, Vice Chair for Research, Department of Medicine, Director, Division of Clinical Immunology and Allergy, Chief, Laboratory of Behavioral Immunology Research, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2012-0255
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Elderly Immune Senescence
Keywords: Immulina; Elderly; Immune
MeSH Terms: interventions — Immulina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator): 10 participants will be randomized to take 1 capsule of placebo daily.
  Interventions: Dietary Supplement: Immulina
- Immulina 200 mg/day (Experimental): 10 participants will be randomized to take 200 mg/day of Immulina.
  Interventions: Dietary Supplement: Immulina
- Immulina 400 mg/day (Experimental): 10 participants will be randomized to take 400 mg/day of Immulina.
  Interventions: Dietary Supplement: Immulina
- Immulina 800 mg/day (Experimental): 10 participants will be randomized to take 800 mg/day of Immulina.
  Interventions: Dietary Supplement: Immulina

INTERVENTIONS:
Dietary Supplement: Immulina
  Other Names: Spirulina

SUMMARY:
This will be a small study aimed at determining the effects of oral Immulina consumption on the immune system in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older;
* Generally otherwise healthy for age and not taking medications/supplements that could be expected to affect stress responses and/or impact immune parameters (example - systemic steroids, beta blockers, antidepressants, anti-anxiety drugs, Echinacea supplements, ginseng supplements or Spirulina supplements).

Exclusion Criteria:

* Inability to comprehend and speak English;
* Any history of major psychological or psychiatric illness (example - dementia, psychotic disorder, acute mania, current substance abuse) that may limit participant cooperation or compromise the integrity of self-reported clinical or psychological data;
* Presence of a confounding underlying systemic illness which could interfere with immunological profiles (example - severe cardiovascular, pulmonary, hepatic, gastrointestinal, renal, neurological, musculoskeletal endocrine , or metabolic systems; other gross physical impairments; or any history of significant convulsive disorder). Specifically, patients with congestive heart failure, recent viral or bacterial illness in the past 3 weeks, chronic kidney disease, thyroid disorder, autoimmune disease will be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Interferon gamma (IFNg) | 8 weeks
  Increase in IFNg from baseline to 8 weeks

SECONDARY OUTCOMES:
Psychological Measures | 8 weeks
  Effects of Immulina on immune biomarkers based upon psychological differences including perceived stress, anxiety, depression and worry
Optimal supplement regime | 8 weeks
  Optimizing Immulina dose for maximal immune biomarker levels observing changes in Treg, Tr1, Th3, T Helper1, T Helper 2 cells, salivary cortisol, salivary alpha amylase, Interleukin 4 and Interleukin 10 cytokine production from baseline to 8 weeks
Demographic differences | 8 weeks
  Effects of Immulina based upon demographic differences including gender, race, age, BMI and socioeconomic status
Immune biomarkers | 8 weeks
  Changes in Treg, Tr1, Th3, T Helper 1, T Helper 2 cells, salivary cortisol, salivary alpha amylase, Interleukin 4 and Interleukin 10 cytokine production from baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D. Marshall, Jr., MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States